CLINICAL TRIAL: NCT06467188
Title: Turkish Validity and Reliability of the Haptotherapeutic Well-Being Scale
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Assist. Prof., Trakya University
Other Study IDs: 14.09.2023-14
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Therapeutic Agalactia
Keywords: Haptonomy; Validity; Reliability; Scale
MeSH Terms: interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validity and reliability — In order to evaluate the content validity of the Turkish version of the scale, 12 expert researchers in the field of gynecology and obstetrics were consulted. The experts were asked to evaluate the items as 1-Not Appropriate, 2-Somewhat Appropriate, 3-Reasonably Appropriate, and 4-Very Appropriate. Experts were asked to suggest items not evaluated as "very appropriate". In the Davis technique, the content validity index which is calculated by dividing the number of experts who marked the options a (The item is appropriate) and b (The item needs minor revision) for each item by the total number of experts providing opinions is expected to be over 0.80 [30]. Based on expert opinions, the content validity index (CVI) value of the scale was calculated to be 96%, meaning that content validity was ensured. The items were reorganized by considering the experts' suggestions. The scale was administered to 252 women over 18 who were included in the study sample after scoring.

SUMMARY:
Objectives: Haptotherapy fosters a sense of unity between the body, mind, and emotions. In addition, it contributes to expanding the woman's perception of her pregnancy and developing a more positive attitude towards pregnancy and childbirth. The study aims to examine the Turkish validity and reliability of the Haptotherapeutic Well-Being Scale, which will be used to evaluate the well-being levels of haptonomy and haptotherapy practices in women.

Design: The study was methodological type. Methods: The study conducted between October 20 and December 20, 2023, with 242 women who volunteered to participate by sharing forum pages on social media (Facebook, Instagram) via the web. Data were collected using a personal information form, including sociodemographic and obstetric characteristics and the Haptotherapeutic Well-Being Scale.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 age, living in Turkiye, using social media (Facebook, Instagram), and agreeing to participate in the study.

Exclusion Criteria:

* Women who were illiterate in Turkish, had hearing-vision problems or mental disabilities, did not have social media (Facebook, Instagram), and did not volunteer to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — over 18 age
Study Population: Women over 18 age, living in Turkiye, using social media (Facebook, Instagram), and agreeing to participate in the study
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Haptotherapeutic Well-Being Scale | 1 day
  Scale consists of 14 items and five sub-dimensions. High scores obtained from the scale mean that the level of haptotherapeutic well-being is also good. There are are received that the minimum 4, maximum 20 points from the psychological well-being sub-dimension, minimum 2, maximum 10 points from the physical health sub-dimension, minimum 3, maximum 15 points from the autonomy, relationships with others and touching and being touched sub-dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kucukkaya B, Isik HK, Rathfisch G. Turkish validity and reliability of the Haptotherapeutic Well-Being Scale. BMC Complement Med Ther. 2024 Aug 30;24(1):323. doi: 10.1186/s12906-024-04613-z. PMID 39215291